CLINICAL TRIAL: NCT04284839
Title: The Direct Oral Anticoagulation Versus Vitamin K Antagonist After Cardiac Surgery Trial
Acronym: DANCE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: DANCE-2020
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Bleeding Post Cardiac Surgery; Indication for Anticoagulation
Keywords: Direct Oral Anticoagulant; Vitamin K Antagonist; Bleeding
MeSH Terms: conditions — Hemorrhage | interventions — apixaban; Dabigatran; edoxaban; Rivaroxaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct Oral Anticoagulation (DOAC) (Active Comparator): Patients in the intervention group will receive a DOAC at doses recommended for the indication, adjusted for their renal function is required. The choice of DOAC will be at the discretion of the treating physician.
  Interventions: Drug: DOAC
- Vitamin K Antagonist (Placebo Comparator): Patients in the control group will receive VKA once daily; the individual dose will be titrated to achieve a guideline-recommended INR range.
  Interventions: Drug: VKA

INTERVENTIONS:
Drug: DOAC — Patients will receive a DOAC at doses recommended for the indication, adjusted for their renal function is required. The choice of DOAC will be at the discretion of the treating physician.
  Other Names: Apixaban; Dabigatran; Edoxaban; Rivaroxaban
  Arms: Direct Oral Anticoagulation (DOAC)
Drug: VKA — Patients in the control group will receive VKA once daily; the individual dose will be titrated to achieve a guideline-recommended INR range.
  Other Names: Warfarin
  Arms: Vitamin K Antagonist

SUMMARY:
The DANCE Trial is a multi-centre, randomized controlled trial comparing the safety of direct oral anticoagulants (DOAC) versus vitamin K antagonists (VKA) in the early period (30 days) after cardiac surgery in patients with atrial fibrillation requiring oral anticoagulation.

DETAILED DESCRIPTION:
Approximately 36,000 Canadian adults undergo cardiac surgery annually. Of these patients, about 10% have a prior history of atrial fibrillation (AF). In the early post-operative period after cardiac surgery, 30-60% of patients develop AF and, by the time of discharge, 32% of patients who underwent cardiac surgery have an indication for oral anticoagulation (OAC). AF is associated with a significantly higher risk of stroke, even when transient, and OAC is the standard for thromboembolic prevention in these patients. In the post-operative period, the balance of benefits and risks of OAC may differ and the safest and most effective OAC in that patient population is uncertain.

Vitamin K antagonists (VKAs), such as warfarin or coumadin, are the most used anticoagulants after cardiac surgery. In the Left Atrial Appendage Occlusion Study (LAAOS) III that recruited 4811 patients from 105 centres in 27 countries, 77% of patients with AF on OAC were discharged on a VKA after cardiac surgery. Among patients taking a DOAC preoperatively, 55% were switched to a VKA after surgery. Over the first post-operative year, most of those patients were gradually transitioned back to a DOAC. Although effective, the use of VKAs is limited by a narrow therapeutic index requiring frequent international normalized ratio (INR) measurements to ensure appropriate levels of anticoagulation. This key limitation leads to non-compliance and discontinuation. In addition, in the first 3 months after cardiac surgery, time in the therapeutic range is low, even with close monitoring by experienced prescribers.

In the last decade, DOACs - inhibitors of factor Xa or thrombin- have become broadly used in patients with AF. Treatment with a DOAC in patients with AF has been demonstrated to yield a lower risk of stroke or systemic embolism and a similar risk of major bleeding when compared to VKAs during long-term follow-up. Moreover, DOACs are more convenient for both patients and clinicians. They have a rapid onset of effect, fixed dosage that obviates the need for regular monitoring, and few interactions with food and other medications. In the postoperative setting, DOACs may also lead to shorter length of stay and reduced costs.

The purpose of this study is to establish whether DOACs are as safe as VKAs in the first few weeks after heart surgery. The results of this study will impact the treatment of hundreds of thousands of patients in the world every year.

A subset of 910 DANCE participants with a recent bioprosthetic aortic and/or mitral valve replacement will be enrolled in the SUNDANCE substudy (Subclinical valve thrombosis in patients with surgical bioprosthetic valve replacement: An imaging substudy of the DANCE trial). SUNDANCE will examine the effects of DOACs versus VKAs on subclinical valve thrombosis and bioprosthetic valve function by conducting computed tomography (CT) scans and echocardiograms at 60 to 90 days after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of enrolment,
2. Open heart surgery in the last 10 days,
3. Atrial fibrillation requiring anticoagulation (including pre-existing or post-operative atrial fibrillation),
4. Informed consent from either the patient or a substitute decision-maker.

Exclusion Criteria:

1. Mechanical valve replacement,
2. Antiphospholipid syndrome (triple positive),
3. Severe renal failure (Cockcroft-Gault equation; creatinine clearance <15 ml/min),
4. Known significant liver disease (Child-Pugh classification B and C),
5. Left ventricular thrombus,
6. Ongoing bleeding, hemorrhagic disorders, or bleeding diathesis,
7. Known contraindication for any DOAC or VKA,
8. Women who are pregnant, breastfeeding, or of childbearing potential,
9. Surgery including left ventricular assist device implantation or cardiac transplantation,
10. Previously enrolled in this trial,
11. Follow-up not possible,
12. History of moderate or severe mitral valvular lesion (stenosis or regurgitation) that is not corrected during index cardiac surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2021-07-18 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Major Bleeding | 30-Days post-randomization
  Major bleeding at 30 days, defined as bleeding that results in death and/or symptomatic bleeding in a critical area or organ, bleeding into a surgical site requiring reoperation, bleeding leading to hospitalization (including presentation to an acute care facility without overnight stay) and/or bleeding that causes a drop in the hemoglobin level of 20g/L or more or that which requires the transfusion of ≥2 units of packed red blood cells or whole blood (as defined by the International Society of Thrombosis and Hemostasis)

SECONDARY OUTCOMES:
Composite of stroke and non-central nervous system systemic arterial embolism at 30 and 90 days. | 30-Days and 90-Days post-randomization
Major Bleeding | 90-Days post-randomization
Pleural or pericardial effusion requiring drainage | 30-Days and 90-Days post-randomization
Systemic arterial embolism | 30-Days and 90-Days post-randomization
Ischemic stroke | 30-Days and 90-Days post-randomization
Deep vein thrombosis | 30-Days and 90-Days post-randomization
Pulmonary Embolism | 30-Days and 90-Days post-randomization
Length of post-operative hospital stay | 30-Days and 90-Days post-randomization
All-Cause Mortality | 6 Months post-randomization

OTHER OUTCOMES:
Minor Bleeding | 30-Days and 90-Days post-randomization
  Tertiary outcome
All bleeding (major plus minor) | 30-Days and 90-Days post-randomization
  Tertiary outcome
Myocardial Infarction | 30-Days and 90-Days post-randomization
Valve Thrombosis | 30-Days and 90-Days post-randomization
  Tertiary outcome
Hemorrhagic stroke | 30-Days and 90-Days post-randomization
  Tertiary outcome
All Stroke | 30-Days and 90-Days post-randomization
  Tertiary outcome
All Arterial Thrombosis/thromboembolism | 30-Days and 90-Days post-randomization
  Tertiary outcome: ischemic stroke, systemic arterial embolism, myocardial infarction, valve thrombosis
Quality of Life - EQ-5D-5L | 30-Days and 90-Days post-randomization
  Tertiary outcome: Measured by The EQ-5D-5L Questionnaire
Patient Satisfaction with Anticoagulant treatment | 30-Days and 90-Days post-randomization
  Tertiary outcome: Assessed by the Perception of Anticoagulant Treatment Questionnaire
Subclinical Valve Thrombosis on CT scan | 60 to 90-Days post-randomization
  Substudy outcome
Mean Aortic Valve g=Gradient on echocardiogram | 60 to 90-Days post-randomization
  Substudy outcome
Aortic Valve Reintervention | 60 to 90-Days post-randomization
  Substudy outcome
Association between subclinical valve thrombosis and clinically significant aortic valve thrombosis, stroke or systemic embolism | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Belley-Cote, MD, MSc, Principal Investigator — McMaster University
Locations (19):
- Australia (2):
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Royal Melbourne Hospital, University of Melbourne, Parkville, Victoria
- Canada (12):
  - University of Alberta Hospital, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Health Science Centre, St. John's, Newfoundland and Labrador
  - Health Sciences North Research Institute, Greater Sudbury, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Hôpital Sacré-Coeur de Montréal, Montreal, Quebec
  - IUCPQ-ULaval, Québec, Quebec
- Germany (5):
  - Heart Center Leipzig, Leipzig, Saxony
  - University Hospital Jena, Jena, Thuringia
  - University Hospital Bonn Heart Center, Bonn
  - West-German Heart and Vascular Center, University of Duisburg-Essen, Essen
  - University Medical Center Hamburg-Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: No
We will establish a plan for the full-scale study but there is no plan to make IPD available to other researchers.